CLINICAL TRIAL: NCT02358317
Title: The Effects of Video Game Learning on the Brain in Adolescents With Autism: A Pilot Study
Brief Title: Motor Learning and Brain Changes in Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-1499
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Autistic Disorder
Keywords: Autism; Postural Stability; Exergaming; White Matter
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video Game Motor Training (Experimental): Participants in the treatment group will come to the University of Wisconsin lab for six weeks to train 3-5 days each week under research staff supervision. Each training session will last 30-60 minutes and will include playing our in-house Ninja Training game combined with balance games from the Wii Fit.
  Interventions: Behavioral: Video Game Motor Training
- Sedentary Video Game Training (Active Comparator): Participants randomly assigned to this condition will come to the lab for six weeks to play sedentary video games 3-5 days each week under research staff supervision. Each training session will last 30-60 minutes. Pre-and post assessments will be done identically to the Experimental group.
  Interventions: Behavioral: Sedentary Video Game Training

INTERVENTIONS:
Behavioral: Video Game Motor Training
  Arms: Video Game Motor Training
Behavioral: Sedentary Video Game Training
  Arms: Sedentary Video Game Training

SUMMARY:
The purpose of this pilot study is to determine whether a video-game based motor training can affect postural stability, daily living skills, autism symptoms, and white matter microstructure of the corticospinal tract in adolescents with Autism Spectrum Disorder (ASD).

DETAILED DESCRIPTION:
Participants: Participants will include 30 adolescents with ASD (13-17 years of age) and 30 adolescents with typical development. Exclusion criteria consists of engaging in more than 2 hours/week of balance training activities (i.e., yoga, tai chi, Wii/Kinect balance games) at study start. Each individual will receive a pre-training magnetic resonance imaging (MRI) scan. Participants will be randomly assigned to either a treatment group or control group. Over the next six weeks, participants in the treatment group will come to the lab to complete 3-5 hours/week of video-game motor training. Participants in the passive control group will come to the lab to do basic motor measurements and sedentary video gaming without motor training. Participants will be asked not to start any new exercise-related programs during those 6 weeks. After the sixth week, all participants will complete a post-training MRI scan and behavioral assessment.

Motor Video Game Training: Participants in the treatment group will come to the University of Wisconsin lab to train 3-5 days each week under research staff supervision. Each training session will last 30-60 minutes and will begin and end with ~5 minutes playing the Ninja Training game from Dr. Ellertson's lab (Boise State University). In this game, participants will hold a position (i.e., the Karate Kid crane pose) for as long as they can, while we collect time-series data on the position of each joint using the Kinect camera as well as time-series data on the center of pressure using the Wii balance board. Participants are rewarded for holding the pose as long as possible by seeing the background behind them come to life. For the rest of the training, participants will play balance games from the Wii Fit.

Motor & Symptom Severity Assessments: Pre-post postural stability measures will be assessed in both groups through standing postures on the Wii balance board (as in Travers et al., 2013). Pre-post symptom severity measures will include parent-report measures of social function, repetitive behaviors/restricted interests, and measures of daily living skills.

Imaging Protocol: Pre- and post-training brain imaging will be completed using a 3 Tesla (ET) MRI scanner with a Nova 32-Channel Head Coil. All scanning will be performed in <60 minutes. Pulse sequences and protocols include advanced diffusion weighted imaging (DWI) with NODDI (Zhang et al., 2012) and multicomponent T1 and T2 relaxometry using steady state sequences (mcDESPOT; Deoni et al., 2008; Alexander et al., 2011). Structural imaging of anatomical detail for morphometric analyses will also be performed using a custom MP2RAGE sequence, which inherently removes the intensity variations from inhomogeneities in the coil sensitivities.

ELIGIBILITY:
Inclusion Criteria for ASD group:

* Previous diagnosis of Autism Spectrum Disorder (ASD)
* Meet criteria for ASD on the Autism Diagnostic Observation Scale (ADOS) and Social Communication Questionnaire (SCQ).

Exclusion Criteria:

* Co-occuring tuberous sclerosis, fragile X, a history of severe head injury, intellectual disability (IQ<70), or hypoxia-ischemia.
* Participants will not be able to be already engaged in more than 2 hours/week of balance training activities (i.e., yoga, tai chi, Wii/Kinect balance games) at study start

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Balance Time | 6 weeks
Postural Stability | 6 weeks
  Center of Pressure Measurements from Wii Balance Board
White matter microstructure of the Corticospinal tract | 6 weeks
  White matter microstructure of the Corticospinal tract, as measured through Diffusion Weighted Imaging

SECONDARY OUTCOMES:
Adaptive Daily Living Skills | 6 weeks
  Vineland-II and Waisman Adaptive Daily Living Skills Measurements
Social Responsiveness | 6 weeks
  Social Responsiveness Scale (SRS) Measurements

CONTACTS AND LOCATIONS:
Overall Officials: Brittany G Travers, Ph.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Waisman Center, University of Wisconsin-Madison, Madison, Wisconsin, United States

REFERENCES:
- [Background] Travers BG, Powell PS, Klinger LG, Klinger MR. Motor difficulties in autism spectrum disorder: linking symptom severity and postural stability. J Autism Dev Disord. 2013 Jul;43(7):1568-83. doi: 10.1007/s10803-012-1702-x. PMID 23132272
- [Background] Deoni SC, Rutt BK, Arun T, Pierpaoli C, Jones DK. Gleaning multicomponent T1 and T2 information from steady-state imaging data. Magn Reson Med. 2008 Dec;60(6):1372-87. doi: 10.1002/mrm.21704. PMID 19025904
- [Background] Alexander AL, Hurley SA, Samsonov AA, Adluru N, Hosseinbor AP, Mossahebi P, Tromp do PM, Zakszewski E, Field AS. Characterization of cerebral white matter properties using quantitative magnetic resonance imaging stains. Brain Connect. 2011;1(6):423-46. doi: 10.1089/brain.2011.0071. Epub 2012 Jan 27. PMID 22432902
- [Background] Zhang H, Schneider T, Wheeler-Kingshott CA, Alexander DC. NODDI: practical in vivo neurite orientation dispersion and density imaging of the human brain. Neuroimage. 2012 Jul 16;61(4):1000-16. doi: 10.1016/j.neuroimage.2012.03.072. Epub 2012 Mar 30. PMID 22484410